CLINICAL TRIAL: NCT00093613
Title: A Phase I Trial of BAY 43-9006 for Patients With Recurrent or Progressive Malignant Glioma
Brief Title: Sorafenib in Treating Patients With Recurrent or Progressive Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03102; NCI-2012-03102 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NABTT-0401; ABTC-0401; NABTT 0401 (Other: Adult Brain Tumor Consortium); NABTT-0401 (Other: CTEP); U01CA062475 (NIH)
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2013-12

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Oligodendroglioma; Adult Giant Cell Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Sorafenib

ARMS (1):
- Treatment (sorafenib tosylate) (Experimental): Patients receive oral sorafenib twice daily on days 1-28 (once daily on day 1 of course 1 only). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients per stratum receive escalating doses of sorafenib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 3 of 6 patients experience dose-limiting toxicity.
  Interventions: Drug: sorafenib tosylate; Other: pharmacological study

INTERVENTIONS:
Drug: sorafenib tosylate — Given PO
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of sorafenib in treating patients with recurrent or progressive malignant glioma. Sorafenib may stop the growth of tumor cells by stopping blood flow to the tumor and by blocking the enzymes necessary for their growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of BAY 43-9006 when administered to adults with recurrent malignant glioma, receiving (Group A) or not receiving (Group B) anticonvulsants known to be metabolized by the P450 hepatic enzyme complex.

II. To assess and estimate the dose-related toxicities. III. To describe the pharmacokinetics of this route of administration, measuring BAY 43-9006, and to assess the pharmacokinetic difference between patients taking enzyme-inducing agents and those who are not.

IV. To estimate overall survival.

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified according to the concurrent use of cytochrome P450-inducing anticonvulsants (yes vs no).

Patients receive oral sorafenib twice daily on days 1-28 (once daily on day 1 of course 1 only). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients per stratum receive escalating doses of sorafenib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 3 of 6 patients experience dose-limiting toxicity.

Patients are followed every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven malignant glioma (anaplastic astrocytoma, anaplastic oligodendroglioma or glioblastoma multiforme) which is progressive or recurrent after radiation therapy ± chemotherapy; patients with previous low grade glioma who progressed after radiotherapy ± chemotherapy and are biopsied and found to have a high grade glioma are eligible
* Patients must have measurable progressive or recurrent malignant glioma by MRI or CT imaging; (Within 14 days before starting treatment)
* Patients must have recovered from toxicity of prior therapy; an interval of at least 3 months must have elapsed since the completion of the most recent course of radiation therapy, while at least 3 weeks must have elapsed since the completion of a non-nitrosourea containing chemotherapy regimen, and at least 6 weeks since the completion of a nitrosourea containing chemotherapy regimen
* Patients must have a Karnofsky performance status >= 60% (i.e. the patient must be able to care for himself/herself with occasional help from others)
* Absolute Neutrophil Count >= 1500/mm^3
* Platelets >= 100,000/mm^3
* Creatinine =< 1.7mg/dl
* Total Bilirubin =< 1.5mg/dl
* Transaminases =< 4 times above the upper limits of the institutional norm
* PT, PTT, INR within institutional norm
* Patients must be able to provide written informed consent
* Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception; women of childbearing potential must have a negative serum pregnancy test; (The anti-proliferative activity of this experimental drug may be harmful to the developing fetus or nursing infant)
* Patients must have a Mini Mental State Exam score >= 15

Exclusion Criteria:

* Patients with serious concurrent infection or medical illness which would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety; (Examples of medical illnesses are [but not limited to] the following: uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements)
* Patients who are pregnant or breast-feeding; (The anti-proliferative activity of this experimental drug may be harmful to the developing fetus or nursing infant)
* Patients who have received more than two prior treatments
* Patients receiving concurrent therapy for their tumor (with the exception of steroids)
* Patients with a concurrent malignancy are ineligible unless they are patients with curatively treated carcinoma-in-situ or basal cell carcinoma of the skin; patients with a prior malignancy are ineligible unless they have been free of disease for >= five years
* Patients must not have any evidence of bleeding diathesis
* Patients must not be on therapeutic anticoagulation; prophylactic anticoagulation (i.e. low dose warfarin) of venous or arterial access devices is allowed provided that the requirements for PT, INR or PTT are met; (Patients will be taken off treatment if they require therapeutic anticoagulation during BAY 43-9006 treatment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2004-12; Primary Completion 2010-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of sorafenib tosylate in patients with recurrent or progressive malignant glioma, receiving (group A) or not receiving (group B) anticonvulsants known to be metabolized by the P450 hepatic enzyme complex | 28 days

SECONDARY OUTCOMES:
Frequency of the toxicities associated with sorafenib tosylate treatment between patients with recurrent or progressive malignant glioma, receiving or not receiving anticonvulsants | Up to 6 years
  The proportion of patients with serious or life threatening toxicities will be estimated along with 95% confidence intervals.
Effect of taking enzyme inducing anticonvulsant drugs on the pharmacokinetics and metabolism of sorafenib tosylate | Days 1 and 15 of course 1 and day 15 of course 2
  The geometric mean +/- standard deviation of the estimated values of the pharmacokinetic parameter for groups of patients evaluated at each dose level will be calculated. Parametric statistical tests (ie, single factor ANOVA, Student's t-test) of pharmacokinetic variables will be performed after logarithmic transformation of the data. All tests will be two-sided and a value of P < 0.05 will be used as the criteria for significance.
Magnitude of variability in the steady-state pharmacokinetics of the drug both within and between patients | Days 1 and 15 of course 1 and day 15 of course 2
  The geometric mean +/- standard deviation of the estimated values of the pharmacokinetic parameter for groups of patients evaluated at each dose level will be calculated. Parametric statistical tests (ie, single factor ANOVA, Student's t-test) of pharmacokinetic variables will be performed after logarithmic transformation of the data. All tests will be two-sided and a value of P < 0.05 will be used as the criteria for significance.
Overall survival | From the time of first day of treatment to death occurrence, assessed up to 6 years
  Non-parametric estimates of survival will be calculated. An overall failure rate will be estimated along with the 95% confidence interval. The overall failure rate is expressed as hazard of failure per person-year of follow-up (the number of deaths divided by the total exposure time in the study cohort).

CONTACTS AND LOCATIONS:
Overall Officials: Louis Nabors, Principal Investigator — National Cancer Institute (NCI)
Locations (10):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Adult Brain Tumor Consortium, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania